CLINICAL TRIAL: NCT06449703
Title: A Randomized, Open-label, Two-period, Cross-over Trial to Evaluate the Single Dose Pharmacokinetics of Insulin Degludec/Liraglutide Injection Compared With Xultophy® in Healthy Chinese Subjects
Brief Title: A Trial to Investigate the Single Dose Pharmacokinetics of Insulin Degludec/Liraglutide in Healthy Chinese Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THDB0213L01
Record Dates: First submitted 2024-06-02; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — IDegLira; Xultophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Degludec/Liraglutide (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Xultophy® (Active Comparator)
  Interventions: Drug: Xultophy®

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Insulin Degludec/Liraglutide combination product with 0.61 mg Liraglutide and 17 U Insulin Degludec, single dose administration under the skin in the abdomen.
  Arms: Insulin Degludec/Liraglutide
Drug: Xultophy® — Xultophy®
  Arms: Xultophy®

SUMMARY:
The main purpose of the trial is to compare the pharmacokinetics of insulin degludec and liraglutide as part of a combination product insulin degludec/liraglutide compared with Xultophy®. During the trial period, serials of blood samples will be collected from the participants at two dosing periods, in order to determine the concentration of insulin degludec and liraglutide. The total volume of blood taken throughout the whole trial period will be less than 400 mL. Participants will be asked to stay on daytime and overnight in the trial sites on some predefined days. For other outpatient days, participants need to attend the trial site as required for drug administration or required assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects signed and dated Informed consent form (ICF) before having a full understanding of the study contents and procedures and potential adverse reactions for the study;
2. Subjects are able to communicate well with the investigator and complete the study;
3. Subjects (including partners) have no pregnancy plan and voluntarily take effective contraceptive measures (For details of the contraceptive measures, see Appendix II) from screening to within 6 months after the last dose of study drug;
4. Healthy Chinese subjects aged 18 to 45 years (inclusive), male or female;
5. Body Mass Index (BMI) ≥ 19 kg/m2 and ≤ 26kg/m2 at screening, male weight ≥ 50 kg, females weight≥ 45 kg;
6. Fasting blood glucose < 6.1 mmol/L at screening;
7. Normal or abnormal but not clinically significant physical examination and vital signs at screening.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. A history of allergy to the ingredients of investigational medical product or other glucagon-like peptide-1 (GLP-1) analogues and their excipients, or a history of severe drug or food allergy;
2. A history of fainting during acupuncture treatment and blood phobia and physical condition unable to withstand blood collection, poor vein condition leading to infeasibility of establishment of blood collection pathway, and difficulty in venous blood collection;
3. Females breast-feeding, or females with a positive blood pregnancy test result at screening;
4. Individuals who have participated in clinical trials of drugs or medical devices within 3 months prior to screening, defined as whose who have used other investigational products or devices;
5. Individuals who have undergone surgery within 3 months prior to screening, which may affect the safety of subjects or the evaluation of the study results as judged by the investigator, or those who have undergone surgery within 1 month prior to screening or plan to undergo surgery during the study;
6. Donated > 400 mL of blood or donated any blood component or had a total blood loss of > 400 mL for any reason within 3 months prior to screening, or those who have a history of blood transfusion, use of blood products or who cannot guarantee not donating whole blood or blood components (e.g., plasma, platelets) during the study or within 30 days after the end of the study;
7. Abnormal and clinically significant clinical laboratory test results, or with the following clinically significant diseases as indicated by other clinical findings within 12 months prior to screening, including but not limited to circulatory, digestion, respiratory, endocrine, urinary, nervous, blood and immune system disorders or psychiatric disorders;
8. A history of diabetes mellitus in the past;
9. A personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2;
10. A history of pancreatitis (acute or chronic) in the past;
11. Thrombotic diseases in the past (e.g., with a medical history of pulmonary embolism and deep venous thrombosis or superficial vein thrombosis not cured or cured within 6 months prior to enrollment) or currently with new thrombotic diseases or using anticoagulants;
12. Abnormal and clinically significant 12-Lead ECG;
13. Abnormal and clinically significant calcitonin test at screening;
14. Positive for any of human immunodeficiency virus (HIV) antibody, hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCVAb) or treponema pallidum antibody;
15. A history of drug abuse in the past 5 years or have engaged in drug taking or been tested positive for breath alcohol test or urine drug screening within 3 months prior to screening;
16. A history of smoking (average daily smoking>5 cigarettes) within 3 months prior to screening and cannot quit during the study;
17. In the three months before screening, the intake of alcohol more than 14 units every week (1 unit ≈ 360 mL of beer, 45 mL of spirits with alcohol content ≥ 40% or 150 mL of wine) and cannot quit during the study;
18. Those who drink excessive amounts of tea, coffee and/or caffeinated beverages (over 8 cups, with 1 cup ≈ 250 mL) every day within 3 months prior to screening and cannot quit during the study;
19. Individuals who have used any prescription drug, non-prescription drug (except for occasional or restrictive use of paracetamol), health product (except for conventional vitamin supplements and calcium) within 14 days prior to screening, or those who have used any traditional herb containing unknown or unspecified components within 3 months prior to screening;
20. Individuals who have received any GLP-1 drug within 3 months prior to screening;
21. Individuals who have received any vaccination within 1 month prior to screening, or plan to receive any vaccination during the study;
22. Individuals who still need or plan to engage in strenuous physical activities or exercise during participation in the study;
23. Any other factor not suitable for participation in this clinical study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-06-16 (Estimated); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma insulin degludec concentration | 0 hours to 120 hours
  Calculated based on insulin degludec measured in plasma
Maximum observed plasma liraglutide concentration | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Area under the plasma insulin degludec concentration time curve | From 0 to last quantifiable observation after single dose of insulin degludec/liraglutide, assessments from 0 hours to 120 hours
  Calculated based on insulin degludec concentration in plasma
Area under the plasma liraglutide concentration time curve | From 0 to last quantifiable observation after single dose of insulin degludec/liraglutide, assessments from 0 hours to 72 hours
  Calculated based on liraglutide concentration in plasma
Area under the plasma insulin degludec concentration time curve from 0 to infinity after single dose | 0 hours to 120 hours
  Calculated based on insulin degludec measured in plasma
Area under the plasma liraglutide concentration time curve from 0 to infinity after single dose | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma

SECONDARY OUTCOMES:
Time to maximum plasma insulin degludec concentration | 0 hours to 120 hours
  Calculated based on insulin degludec measured in plasma
Time to maximum plasma liraglutide concentration | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Terminal elimination half-life for insulin degludec | 0 hours to 120 hours
  Calculated based on insulin degludec measured in plasma
Terminal elimination half-life for liraglutide | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Apparent clearance for insulin degludec | 0 hours to 120 hours
  Calculated based on insulin degludec measured in plasma
Apparent clearance for liraglutide | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Apparent volume of distribution for insulin degludec | 0 hours to 120 hours
  Calculated based on insulin degludec measured in plasma
Apparent volume of distribution for liraglutide | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Area under the plasma insulin degludec concentration time curve | 0 hours to 24 hours
  Calculated based on insulin degludec concentration in plasma
Number of treatment emergent adverse events | From the first drug administration to the follow-up visit (6 to 13 days after the last drug administration)
  Count
Number of treatment emergent hypoglycaemic episodes | From the first drug administration to the follow-up visit (6 to 13 days after the last drug administration)
  Count
Number of participants with injection site reactions (spontaneous pain, tenderness, itching, redness, edema, induration/infiltration) | From the first drug administration to the follow-up visit (6 to 13 days after the last drug administration)
  Count

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Jilin, China

IPD SHARING:
Plan to Share IPD: No